CLINICAL TRIAL: NCT01016041
Title: A Randomized Controlled Trial of Everolimus-eluting Stents and Paclitaxel-eluting Stents for Coronary Revascularization in Daily Practice: The COMPARE Trial
Brief Title: A Trial of Everolimus-eluting Stents and Paclitaxel-eluting Stents for Coronary Revascularization in Daily Practice: The COMPARE Trial
Acronym: COMPARE 1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Maasstad Hospital (Other)
Responsible Party: Pieter Smits, Maasstad Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NL15206.101.06
Record Dates: First submitted 2009-11-16; First posted 2009-11-18 (Estimated); Last update posted 2015-12-28 (Estimated); Status verified 2015-12

CONDITIONS: Stable Angina; Unstable Angina; Acute Coronary Syndrome
Keywords: drug-eluting stent; stable angina; ACS; MACE; safety; stent thrombosis
MeSH Terms: conditions — Angina, Stable; Angina, Unstable; Acute Coronary Syndrome

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- everolimus stent (Experimental)
  Interventions: Device: everolimus stent
- paclitaxel eluting (Active Comparator)
  Interventions: Device: paclitaxel stent

INTERVENTIONS:
Device: everolimus stent — stenting
  Arms: everolimus stent
Device: paclitaxel stent — stenting
  Arms: paclitaxel eluting

SUMMARY:
Instead of treating in-stent restenosis, the best strategy for patients is preventing in-stent restenosis. Recent advances in the understanding of the cellular mechanism responsible for smooth muscle cell proliferation (neointimal hyperplasia), together with improvement in stent coating and eluting technology have provided the scientific background to develop drug eluting stents. Drug eluting stents (DES) are now the most promising development in interventional cardiology. Different classes of drugs mounted in a polymer layer on the surface of the stent have shown to be very effective in preventing neointimal hyperplasia. Currently there are 7 DES stents CE marked and commercially available on the market. Two stents, respectively the sirolimus eluting Cypher™ stent and the paclitaxel eluting Taxus™ stent, are in clinical use since 2002. The Cypher™ stent consists of the Bx sonic stent/balloon platform. The stent is coated with a non-degradable biocompatible PBMA/PEVA polymer which elutes sirolimius. The Taxus™ stent consists of the Express2 balloon/stent platform coated with non-degradable biocompatible Translute™ polymer which elutes paclitaxel.

Recent large randomized trials like RAVEL, SIRIUS, E-SIRIUS C-SIRIUS (Cypher™ versus bare metal BX sonic™ stent), TAXUS II, IV, V, VI (Taxus versus bare metal Express™ stent) have shown that DES dramatically reduce the incidence of in-stent restenosis and subsequently the need for target lesion revascularization in patients with non complex and moderate long de-novo coronary lesions in vessels with a diameter between 2.5 -3.5 mm.1-11 Considering the very encouraging results of these early clinical trials with so far mid long term follow-up, there is the need to explore the utilization of DES in the other subsets of coronary lesions like: long lesions, chronic total occlusions, venous graft lesions, thrombotic lesions, restenosis lesions, ostial and bifurcation lesions and lesions in large vessels.

As the result from the previous reported randomized trials, FDA and other regulatory institutes require that new DES are now being evaluated against one of the former DES (Cypher or Taxus). The XIENCE-V stent is a second generation DES, with thinner and more flexible Cobalt-Chromium stent struts, compared to the first generation Stainless Steel stent struts of Cypher and Taxus. This study addresses the questions whether the XIENCE-V™ stent has superior clinical results as the Taxus™ stent in the general population that is being referred for percutaneous coronary intervention (PCI).

Objective of the study:

The main objective of the study is a head tot head comparison of the everolimus coated XIENCE-V™ stent with the paclitaxel coated TAXUS™ stent in order to observe whether there is a difference in clinical outcome between both stents.

Efficacy of both stents will be assessed by the composite end point of: all death, non fatal myocardial infarction and target vessel revascularization.

Study design:

Single center, randomised, open label study in all-comers referred for PCI.

Study population:

Approximately 1600 consecutive patients with coronary artery disease who are eligible according to the in- and exclusion criteria will be enrolled and randomized on a 1:1 basis.

Primary study parameters/outcome of the study:

The primary end point of the study is the composite end point of: all death, non fatal myocardial infarction, target vessel revascularization at 1 year.

Secondary study parameters/outcome of the study:

The secondary end points of the study are:

A) The combined endpoint of cardiac death, non fatal myocardial infarction, ischemic driven target lesion revascularization (TLR) rate at 1, 6 and 12 months follow-up.

B) The combined endpoint of all death, non fatal myocardial infarction, target vessel revascularization (TVR) rate at 2, 3, 4 and 5 years.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness:

The burden for the patient consists of filling in 8 questionnaires (1 A4 per questionnaire) in 5 years time.

The first 3 questionnaires in the first year are also requested for monitoring purposes by the Ministry of Health and the Dutch Cardiology Society (Nederlandse Vereniging Voor Cardiologie; NVVC).

There is no risk for the patient related to participation in this study. The patient will receive a Taxus or Xience-V stent anyhow, if the indication for a DES stent exists.

ELIGIBILITY:
Inclusion Criteria:

* Any patient from 18 to 85 years with lesions feasible for PCI treatment.

Exclusion Criteria:

* Dual antiplatelet therapy contraindication,
* Participation in other trials,
* No informed consent.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1800 (Actual)
Dates: Start 2007-02; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
The primary end point of the study is the composite end point of: all death, non fatal myocardial infarction, target vessel revascularization at 1 year. | 1 year

SECONDARY OUTCOMES:
The combined endpoint of cardiac death, non fatal myocardial infarction, ischemic driven target lesion revascularization (TLR) rate at 1, 6 and 12 months follow-up. | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Maasstad Hospital, Rotterdam, Netherlands

REFERENCES:
- [Derived] Smits PC, Vlachojannis GJ, McFadden EP, Royaards KJ, Wassing J, Joesoef KS, van Mieghem C, van de Ent M. Final 5-Year Follow-Up of a Randomized Controlled Trial of Everolimus- and Paclitaxel-Eluting Stents for Coronary Revascularization in Daily Practice: The COMPARE Trial (A Trial of Everolimus-Eluting Stents and Paclitaxel Stents for Coronary Revascularization in Daily Practice). JACC Cardiovasc Interv. 2015 Aug 17;8(9):1157-1165. doi: 10.1016/j.jcin.2015.03.028. Epub 2015 Jul 22. PMID 26210806
- [Derived] Claessen BE, Smits PC, Kereiakes DJ, Parise H, Fahy M, Kedhi E, Serruys PW, Lansky AJ, Cristea E, Sudhir K, Sood P, Simonton CA, Stone GW. Impact of lesion length and vessel size on clinical outcomes after percutaneous coronary intervention with everolimus- versus paclitaxel-eluting stents pooled analysis from the SPIRIT (Clinical Evaluation of the XIENCE V Everolimus Eluting Coronary Stent System) and COMPARE (Second-generation everolimus-eluting and paclitaxel-eluting stents in real-life practice) Randomized Trials. JACC Cardiovasc Interv. 2011 Nov;4(11):1209-15. doi: 10.1016/j.jcin.2011.07.016. PMID 22115661
- [Derived] Planer D, Smits PC, Kereiakes DJ, Kedhi E, Fahy M, Xu K, Serruys PW, Stone GW. Comparison of everolimus- and paclitaxel-eluting stents in patients with acute and stable coronary syndromes: pooled results from the SPIRIT (A Clinical Evaluation of the XIENCE V Everolimus Eluting Coronary Stent System) and COMPARE (A Trial of Everolimus-Eluting Stents and Paclitaxel-Eluting Stents for Coronary Revascularization in Daily Practice) Trials. JACC Cardiovasc Interv. 2011 Oct;4(10):1104-15. doi: 10.1016/j.jcin.2011.06.018. PMID 22017936
- [Derived] Stone GW, Rizvi A, Sudhir K, Newman W, Applegate RJ, Cannon LA, Maddux JT, Cutlip DE, Simonton CA, Sood P, Kereiakes DJ; SPIRIT IV Investigators. Randomized comparison of everolimus- and paclitaxel-eluting stents. 2-year follow-up from the SPIRIT (Clinical Evaluation of the XIENCE V Everolimus Eluting Coronary Stent System) IV trial. J Am Coll Cardiol. 2011 Jun 28;58(1):19-25. doi: 10.1016/j.jacc.2011.02.022. Epub 2011 Apr 21. PMID 21514084
- [Derived] Smits PC, Kedhi E, Royaards KJ, Joesoef KS, Wassing J, Rademaker-Havinga TA, McFadden E. 2-year follow-up of a randomized controlled trial of everolimus- and paclitaxel-eluting stents for coronary revascularization in daily practice. COMPARE (Comparison of the everolimus eluting XIENCE-V stent with the paclitaxel eluting TAXUS LIBERTE stent in all-comers: a randomized open label trial). J Am Coll Cardiol. 2011 Jun 28;58(1):11-8. doi: 10.1016/j.jacc.2011.02.023. Epub 2011 Apr 21. PMID 21514083
- [Derived] Kedhi E, Joesoef KS, McFadden E, Wassing J, van Mieghem C, Goedhart D, Smits PC. Second-generation everolimus-eluting and paclitaxel-eluting stents in real-life practice (COMPARE): a randomised trial. Lancet. 2010 Jan 16;375(9710):201-9. doi: 10.1016/S0140-6736(09)62127-9. Epub 2010 Jan 7. PMID 20060578